CLINICAL TRIAL: NCT00632138
Title: MAPS (Men After Prostate Surgery) : Conservative Treatment for Men With Urinary Incontinence After Prostate Surgery; Multicentre Randomised Controlled Trial of Pelvic Floor Muscle Training and Biofeedback [MAPS]
Brief Title: Pelvic Floor Muscle Training and Biofeedback or Standard Therapy in Men Who Have Undergone Radical Prostatectomy or Transurethral Resection of the Prostate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aberdeen Royal Infirmary (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: ABROIN-MAPS; CDR0000586420 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN87696430; NCT00237029 (obsolete NCT alias)
Record Dates: First submitted 2008-03-07; First posted 2008-03-10 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-12

CONDITIONS: Nonmalignant Neoplasm; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Sexual Dysfunction; Urinary Incontinence
Keywords: sexual dysfunction; psychosocial effects of cancer and its treatment; prostate cancer; benign prostatic hyperplasia; urinary incontinence
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Sexual Dysfunction, Physiological; Urinary Incontinence; Prostatic Hyperplasia | interventions — Biofeedback, Psychology; Psychiatric Rehabilitation

INTERVENTIONS:
Behavioral: exercise intervention
Other: questionnaire administration
Procedure: biofeedback
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Personalized training by a health professional may improve urinary incontinence. It is not yet known whether pelvic floor muscle training and biofeedback are more effective than standard therapy in improving urinary continence after radical prostatectomy or transurethral resection of the prostate.

PURPOSE: This randomized phase III trial is studying pelvic floor muscle training and biofeedback to see how well it works compared with standard therapy in men who have undergone radical prostatectomy or transurethral resection.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish whether conservative physical treatment delivered personally by a trained health professional results in better urinary and other outcomes compared with standard management in men who are incontinence after prostate surgery.

OUTLINE: This is a multicenter study. Patients are stratified according to type of operation (radical prostatectomy vs transurethral resection of prostate). Patients are randomized to 1 of 2 treatment arms.

* Arm I (intervention group): At 6 weeks after surgery, patients undergo an assessment of their symptoms by a physiotherapist or continence nurse. All patients are taught pelvic floor muscle training and men with urgency or urge incontinence are also taught bladder training. Pelvic floor training consists of 3 maximum pelvic floor contractions in 3 positions (standing, sitting, and lying down) twice a day, lifting of the pelvic floor while walking, tightening of the pelvic muscles before activities, and tightening of the pelvic muscles after urinating to squeeze out any last drops. The strength of the pelvic floor contractions is monitored by biofeedback involving digital anal assessment and relaying the information back to men in order that they know when they are performing contractions correctly and to inform them when they are increasing the strength or duration of their contractions. Therapists may use machine-mediated biofeedback with an anal biofeedback probe at their discretion in addition to digital anal assessment. Bladder training consists of gradually delaying urination by pelvic floor muscle contraction and distracting activities to teach the bladder to hold increasing volumes of urine. Patients also receive a customized Pelvic Floor Exercise Booklet describing pelvic floor muscle training in addition to a customized Lifestyle Advice Booklet giving general lifestyle advice. Patients have reinforcement sessions at approximately 2, 6, and 12 weeks after the first appointment.
* Arm II (control group): Patients receive a customized Lifestyle Advice Booklet containing supportive lifestyle advice only (without reference to pelvic floor muscle training) by mail following randomization. Patients do not receive formal assessment or treatment but will be able to access usual care and routine NHS services if they feel they need help, including written advice if this is part of routine hospital care.

All patients keep a urinary diary at 3, 6, 9, and 12 months that includes frequency of urination (day and night), daily episodes of incontinence and quantity of loss, daily use of pads, and the need to change clothing or bedding. A Health Care Utilization Questionnaire will be obtained at 3 and 9 months. Additional questionnaires are obtained at baseline and 6 and 12 months.

The use of NHS services, pads, and practice of pelvic floor muscle training is documented in both groups using information from questionnaires and Urinary Diaries.

Six months after the last patient has been recruited, a check for Scottish men only is performed to compare self-reported operations, diagnoses, and hospital admissions with centrally collected data to validate a proportion of the data.

After completion of study treatment, patients are followed at 6 and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Men who have undergone a radical prostatectomy for prostate cancer or men who have undergone a transurethral resection of the prostate for benign prostatic hypertrophy
* Urinary incontinence at six weeks after prostate surgery

  * Incontinence is defined as a response on the screening questionnaire indicating a loss of urine including how often and how much

PATIENT CHARACTERISTICS:

* Able to comply with intervention
* Able to complete study questionnaires

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No referral for formal therapy (teaching of pelvic floor muscle training) due to prostate surgery
* No concurrent or planned radiotherapy during the first 3 months after surgery
* No palliative endoscopic resection of prostate due to outflow obstruction for advanced prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Subjective report of urinary continence at 12 months
Incremental cost per quality-adjusted year

SECONDARY OUTCOMES:
Subjective report of continence or improvement of urinary incontinence at 3, 6, and 9 months after randomization and improvement at 12 months
Objective report of the number of incontinent episodes in the previous week from the urinary diary
Duration of incontinence based on time of resolution relative to time of operation and randomization
Use of absorbent pads, penile collecting sheath, bladder catheter, or bed/chair pads
Number and type of incontinence products used
Co-existence, cure or development of urgency, or urge incontinence
Urinary frequency
Nocturia
Fecal incontinence (passive or urge)
Other bowel dysfunction (i.e., urgency, constipation, or other bowel diseases)
Sexual function at 12 months including information about erection, ejaculation, retrograde ejaculation, pain, change in sex life, and reason for change
Incontinence-specific quality of life outcome measure using the 10-point scale and ICI questionnaire
General health measures
Need for alternative management for incontinence (e.g., surgery or drugs)
Use of GP, nurse, consultant urologist, or physiotherapist
Visits to GP
Visits to practice nurse
Use of pelvic floor muscle training
Lifestyle changes (i.e., weight, constipation, lifting, coughing, or exercise)
Patient costs (e.g., self care [e.g., pads or laundry], travel to health services, or sick leave)
Cost of conservative trial treatment
Cost of alternative or additional NHS treatments (e.g., pads, catheters, drugs [e.g., adrenergic agonists, anticholinergics, or oral medication for erectile dysfunction], hospital admissions, or further surgery)
Other measures of cost-effectiveness (e.g., incremental cost per additional man continent at 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Cathryn Glazener, MD, Study Chair — Aberdeen Royal Infirmary
Locations (37):
- United Kingdom (37):
  - Tameside General Hospital, Ashton-under-Lyne, England
  - Southmead Hospital, Bristol, England
  - Bristol Royal Infirmary, Bristol, England
  - Mid Cheshire Hospitals Trust- Leighton Hopsital, Crewe, England
  - Royal Bolton Hospital, Farnworth, England
  - King George Hospital, Ilford, Essex, England
  - Ipswich Hospital, Ipswich, England
  - Airedale General Hospital, Keighley, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - St. Mary's Hospital, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - James Cook University Hospital, Middlesbrough, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital, Nottingham, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Queens Hospital, Romford, England
  - Hope Hospital, Salford, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Lister Hospital, Stevenage, England
  - Stepping Hill Hospital, Stockport, England
  - Taunton and Somerset Hospital, Taunton, England
  - Hillingdon Hospital, Uxbridge, England
  - New Cross Hospital, Wolverhampton, England
  - Yeovil District Hospital, Yeovil, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ayr Hospital, Ayr, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Queen Margaret Hospital - Dunfermline, Dunfermline, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Inverclyde Royal Hospital, Greenock, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Morriston Hospital NHS Trust, West Glamorgen, Scotland
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Derived] Johnson EE, Mamoulakis C, Stoniute A, Omar MI, Sinha S. Conservative interventions for managing urinary incontinence after prostate surgery. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD014799. doi: 10.1002/14651858.CD014799.pub2. PMID 37070660